CLINICAL TRIAL: NCT05171881
Title: Brain Oxygenation in Extremely Preterm Infants-II
Brief Title: Brain Oxygenation-II
Acronym: BOx-II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Valerie Chock, M.D., M.S. Epi (Other)
Collaborators: Washington University School of Medicine (Other); Cerebral Palsy Alliance (Other)
Responsible Party: Sponsor-Investigator, Valerie Chock, M.D., M.S. Epi, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 56759b
Record Dates: First submitted 2021-11-26; First posted 2021-12-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Hypoxia
MeSH Terms: conditions — Hypoxia, Brain | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Single arm interventional study to maintain cerebral oxygen saturation in targeted range
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): All infants will undergo non-invasive NIRS monitoring of cerebral oxygen saturation and will have algorithm-driven clinical interventions to maintain cerebral saturation within target range during the first 72 hours of life.
  Interventions: Other: Intervention for cerebral hypoxia

INTERVENTIONS:
Other: Intervention for cerebral hypoxia — For cerebral oxygen saturation measures below target range (cerebral hypoxia), a treatment algorithm with the following potential clinical interventions will be applied: fluid resuscitation, initiation of vasopressor/inotrope medication, change in mechanical ventilation or respiratory support, adjustment of fractional inspired oxygen, transfusion of red blood cells, acquisition of echocardiogram or cranial ultrasound.

SUMMARY:
The Brain Oxygenation-II study (BOx-II) is a phase-II, multicenter, single-arm clinical trial evaluating interventions based on near-infrared spectroscopy (NIRS) monitoring of cerebral oxygen saturation in extremely premature infants. Enrolled infants will follow a treatment guideline to maintain cerebral oxygen saturation in a target range within the first 72 hours of life. The primary outcomes will include interventions used to maintain cerebral saturation in target range, rates of cerebral hypoxia and systemic hypoxia, and a composite of death or severe brain injury detected on term-equivalent magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with postmenstrual age less than 28 weeks
* Signed informed consent

Exclusion Criteria:

* Missing written parental informed consent
* Decision not to conduct full intensive care support
* No possibility to place cerebral NIRS oximeter within six hours after birth
* Skin integrity insufficient to allow for sensor placement as deemed by a clinician

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of interventions used to address cerebral hypoxia | From birth until 72 hours of life
  Frequency of specific interventions chosen to address cerebral hypoxia

SECONDARY OUTCOMES:
Rates of cerebral hypoxia and systemic hypoxia | From birth until 72 hours of life
  Rates of cerebral hypoxia as detected by near-infrared spectroscopy (NIRS) monitoring of cerebral oxygen saturation and systemic hypoxia as detected by conventional pulse oximetry monitoring of systemic oxygen saturation
Rates of death or severe brain injury | 36-42 weeks corrected gestational age
  Rates of death or severe brain injury (including intraventricular hemorrhage, white matter injury, cystic periventricular leukomalacia, cerebellar hemorrhage, post-hemorrhagic ventricular dilation, or cerebral atrophy) detected on term-equivalent magnetic resonance imaging performed between 36 and 42 weeks corrected gestational age.

OTHER OUTCOMES:
Rates of other neonatal morbidities | Birth until hospital discharge, an average of 3 months
  Rates of other neonatal morbidities including bronchopulmonary dysplasia, severe retinopathy of prematurity, and/or mortality before neonatal intensive care unit discharge

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Chock, MD, Principal Investigator — Stanford University; Zachary Vesoulis, MD, Principal Investigator — Washington University in Saint Louis
Locations (5):
- United States (5):
  - Loma Linda University, Loma Linda, California
  - Stanford University, Palo Alto, California
  - Washington University in Saint Louis, St Louis, Missouri
  - University of Texas- Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Vesoulis Z, Hopper A, Fairchild K, Zanelli S, Chalak L, Noroozi M, Liu J, Chock V. A phase-II clinical trial of targeted cerebral near infrared spectroscopy using standardized treatment guidelines to improve brain oxygenation in preterm infants (BOx-II): A study protocol. Contemp Clin Trials. 2022 Sep;120:106886. doi: 10.1016/j.cct.2022.106886. Epub 2022 Aug 19. PMID 35995129